CLINICAL TRIAL: NCT07307105
Title: Comparative Effects Of Creative Movement & Play Based Interventions On Motor Skills, Balance And Quality Of Life In Children With Developmental Delay
Brief Title: Comparative Effects Of Creative Movement & Play Based Interventions On Motor Skills
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: khadija liaquat (Other)
Collaborators: Riphah International University (Other)
Responsible Party: Sponsor-Investigator, khadija liaquat, senior lecturer, Riphah International University
Organization: Riphah International University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Riphah IU Yashma
Record Dates: First submitted 2025-12-14; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Developmental Delay
Keywords: Balance, Quality of Life, Developmental Delay, Motor Skills
MeSH Terms: conditions — Learning Disabilities | interventions — Play Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Creative Movement intervention group. (Experimental): Group A (Creative Movement) engaged in activities such as a Hello Song for upper limb coordination,
  Interventions: Behavioral: creative movement intervention
- Play-Based intervention group (Experimental): Group B (Play-Based Intervention) included obstacle courses, dual-limb coordination games, story reading, building tasks (blocks/LEGOs), and arts & crafts for fine motor development. Each session concluded with a cool-down, promoting relaxation and emotional regulation
  Interventions: Behavioral: play based intervention

INTERVENTIONS:
Behavioral: creative movement intervention — Group A (Creative Movement) engaged in activities such as a Hello Song for upper limb coordination, strength exercises (Grow Strong segment), locomotor games, yoga with breathing, and music-making with instruments. Each session lasted 60 minutes and was conducted twice weekly for 8 weeks
  Arms: Creative Movement intervention group.
Behavioral: play based intervention — Group B (Play-Based Intervention) included obstacle courses, dual-limb coordination games, story reading, building tasks (blocks/LEGOs), and arts & crafts for fine motor development. Each session concluded with a cool-down, promoting relaxation and emotional regulation
  Arms: Play-Based intervention group

SUMMARY:
Children with developmental delay often face challenges in motor skills, balance, and overall quality of life, requiring interventions that are both effective and engaging. The purpose of this study is to improving these areas and investigating comparative effects of both creative movement and play based intervention that can help identify the most effective approach for enhancing motor abilities, balance, and overall well-being in this population

DETAILED DESCRIPTION:
This randomized clinical trial will assess the effects of Creative Movement and Play-Based Interventions on motor skills, balance, and QoL in children with developmental delays. Data will be collected from special education centers and pediatric rehabilitation clinics. Inclusion criteria will include children aged 5-8 years, both genders, with MMSE >24, Stork Stand >4 seconds, and baseline scores on Pediatric Berg Balance Scale, TGMD-2, BOT-2, and PedsQL. Exclusion criteria will cover neurological or musculoskeletal disorders, uncorrected sensory impairments, behavioral issues like ADHD or autism, and recent surgery or assistive device use. Children with chronic illnesses limiting activity, recent specialized motor training, non-compliance with testing. Participants will be randomly assigned to either a Creative Movement or Play-Based Intervention group. Outcome measures will include the Bruininks-Oseretsky Test of Motor Proficiency, Pediatric Balance Scale, Timed Up and Go Test, and Pediatric Quality of Life Inventory. The data collection procedure systematically organized for two intervention groups: Both groups began each session with a 5-minute baseline warm-up including light aerobic movements, dynamic stretching, and active-assisted ROM exercises. Group A (Creative Movement) engaged in activities such as a Hello Song for upper limb coordination, strength exercises (Grow Strong segment), locomotor games, yoga with breathing, and music-making with instruments. Each session lasted 60 minutes and was conducted twice weekly for 8 weeks. Group B (Play-Based Intervention) included obstacle courses, dual-limb coordination games, story reading, building tasks (blocks/LEGOs), and arts & crafts for fine motor development. Each session concluded with a cool-down, promoting relaxation and emotional regulation. Group A will be Creative Movement Intervention and Group B will be Play-Based Intervention, to study Effects of Creative Movement & Play Based Interventions on MotorSkills, balance and quality of life in Children with Developmental Delay.Data will be analyzed using SPSS version 27 to determine the effectiveness of both interventions in enhancing motor function, balance, and overall quality of life

ELIGIBILITY:
inclusion :

1. Children aged 5-8 years.
2. Both girls and boys .
3. Mini-Mental State Examination (MMSE) score > 24 .
4. Stork Stand Balance Test (both legs) > 4 seconds .
5. Pediatric Berg Balance Scale score ≥ 40 .
6. TGMD-2 GMQ score ≤ 79 (≤ 25th percentile) .
7. BOT-2 Total Motor Composite score ≤ 18th percentile .
8. PedsQL total score ≤ 70

Exclusion :

1. Musculoskeletal Impairments affecting posture.
2. balance.
3. Uncorrected visual or auditory impairments .
4. Behavioral or Attention Disorders that may impair test compliance or affect performance reliability .
5. Recent Surgery or Injury in the past 6 months .
6. Use of Assistive Devices .
7. Chronic Illness Affecting Physical Activity .
8. Participation in specialized motor training in the past 3 months .
9. Inability to follow instructions or complete assessments (TGMD-2, BOT-2, PedsQL).

Ages: 5 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2025-10-26 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
PedsQL. | 8 weeks
  Is a standardized, validated tool designed to measure health-related quality of life (HRQOL) in children and adolescents aged 2-18 years. The Turkish validity and reliability tests of the form were performed by Memik et al. (2008). There are other versions of this data collection tool which were developed for different age groups. There is a Likert type answer scale with five answer options: (0 ¼ never, 1 ¼ seldom, 2 ¼ sometimes, 3 ¼ often, 4 ¼ always). The points which are obtained from the items are calculated and a score between 0 and 100 is linearly obtained (0 ¼ 100, 1 ¼ 75, 2 ¼ 50, 3
  ¼ 25, 4 ¼ 0). A score between 0 and 100 indicates the quality of life score and an increase in the scores means an increase in the quality of life.
Bruininks-Oseretsky Test of Motor Proficiency, Second Edition (BOT-2) for fine and gross Motor Skills | 8 weeks
  Is a widely recognized and reliable tool for evaluating both fine and gross motor skills in children aged 4 to 21 years. The shorter form of the test consists of fourteen subtests, which assess fine motor precision and integration, bilateral coordination, balance, running speed, agility, upper body coordination, and strength. The reliability of all the mentioned items is above 0.70, with overall internal consistency reliability ranging from 0.80 to 0.90, and test-retest reliability reported between 0.80 and 0.87, indicating strong measurement stability. It should be noted that the test validity and reliability were established in a sample of healthy children. The short form includes five fine motor skill tests (Drawing, Lines through Paths-Crooked, Folding Paper, Copying a Square, Copying a Star, Transferring Pennies) and nine gross motor tasks (Jumping in Place-Same Sides Synchronized, Tapping Feet and Fingers-Same Sides Synchronized, Walking Forward on a Line, Standing on

SECONDARY OUTCOMES:
Pediatric Balance Scale PBS for Functional Balance | 8 weeks
  Is an adaptation of the Berg Balance Scale and it is a criterion-referenced test assessing functional balance in children 2 years - 7 years and older. It is a valid and reliable balance tool that assesses for functional balance using 14 tasks which are similar to activities of daily living. Within the tasks, the PBS incorporates the conditions similar to the Romberg, Sharpened Romberg, Functional Reach Test and Standing on One Leg test. These tasks can be scored from 0 to 4 where a high score indicates good performance and the test can be completed in approximately 20 min with the aid of easily accessible equipment e.g., chair, bench, stopwatch etc. The PBS has an interrater reliability of (ICC [3, 2] = 0.90-0.92), test-retest (ICC [2,1] = 0.923), and intra-rater reliability (ICC [2,1] = 0.895-0.998) allowing for adequately identifying children with balance dysfunction

CONTACTS AND LOCATIONS:
Locations (1):
- Rax clinic iqbal town, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No